CLINICAL TRIAL: NCT02852005
Title: A Phase 1 Clinical Trial to Evaluate the Immunogenicity of AIDSVAX B/E Bivalent gp120 Vaccine and MVA/HIV62B in Healthy, HIV-1-Uninfected Adult Participants Who Previously Received MVA/HIV62B in DNA/MVA or MVA/MVA Regimens in HVTN 205
Brief Title: Evaluating the Immunogenicity of the AIDSVAX B/E Vaccine and the MVA/HIV62B Vaccine in Healthy, HIV-1-Uninfected Adults Who Previously Received MVA/HIV62B in DNA/MVA or MVA/MVA Regimens in HVTN 205
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 114; 12035 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: MVA/HIV62B + Placebo (Experimental): Participants who received 3 sequential administrations of MVA/HIV62B in HVTN 205 will receive the MVA/HIV62B vaccine in their left deltoid at Months 0 and 4. They will receive placebo in their right deltoid at Months 0 and 4.
  Interventions: Biological: MVA/HIV62B vaccine; Biological: Placebo
- Group 2: MVA/HIV62B + AIDSVAX B/E (Experimental): Participants who received 3 sequential administrations of MVA/HIV62B in HVTN 205 will receive the MVA/HIV62B vaccine in their left deltoid at Months 0 and 4. They will receive the AIDSVAX B/E vaccine in their right deltoid at Months 0 and 4.
  Interventions: Biological: MVA/HIV62B vaccine; Biological: AIDSVAX B/E vaccine
- Group 3: MVA/HIV62B + Placebo (Experimental): Participants who received 2 sequential priming administrations of JS7 DNA plasmid followed by 2 sequential boost administrations of MVA/HIV62B in HVTN 205 will receive the MVA/HIV62B vaccine in their left deltoid at Months 0 and 4. They will receive placebo in their right deltoid at Months 0 and 4.
  Interventions: Biological: MVA/HIV62B vaccine; Biological: Placebo
- Group 4: MVA/HIV62B + AIDSVAX B/E (Experimental): Participants who received 2 sequential priming administrations of JS7 DNA plasmid followed by 2 sequential boost administrations of MVA/HIV62B in HVTN 205 will receive the MVA/HIV62B vaccine in their left deltoid at Months 0 and 4. They will receive the AIDSVAX B/E vaccine in their right deltoid at Months 0 and 4.
  Interventions: Biological: MVA/HIV62B vaccine; Biological: AIDSVAX B/E vaccine
- Group 5: Placebo + AIDSVAX B/E (Experimental): Participants who received 2 sequential priming administrations of JS7 DNA plasmid followed by 2 sequential boost administrations of MVA/HIV62B in HVTN 205 will receive placebo in their left deltoid at Months 0 and 4. They will receive the AIDSVAX B/E vaccine in their right deltoid at Months 0 and 4.
  Interventions: Biological: AIDSVAX B/E vaccine; Biological: Placebo

INTERVENTIONS:
Biological: MVA/HIV62B vaccine — 1×10^8 TCID50 dose to be administered as a 1 mL intramuscular (IM) injection in the deltoid
  Arms: Group 1: MVA/HIV62B + Placebo; Group 2: MVA/HIV62B + AIDSVAX B/E; Group 3: MVA/HIV62B + Placebo; Group 4: MVA/HIV62B + AIDSVAX B/E
Biological: AIDSVAX B/E vaccine — 600 mcg/mL dose to be administered as a 1 mL IM injection in the deltoid
  Arms: Group 2: MVA/HIV62B + AIDSVAX B/E; Group 4: MVA/HIV62B + AIDSVAX B/E; Group 5: Placebo + AIDSVAX B/E
Biological: Placebo — Sodium Chloride for Injection USP, 0.9% to be administered as a 1 mL IM injection in the deltoid
  Arms: Group 1: MVA/HIV62B + Placebo; Group 3: MVA/HIV62B + Placebo; Group 5: Placebo + AIDSVAX B/E

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of the AIDSVAX B/E vaccine and the MVA/HIV62B vaccine in healthy, HIV-1-uninfected adults who previously received MVA/HIV62B in DNA/MVA or MVA/MVA vaccine regimens in the HVTN 205 study.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity of the AIDSVAX B/E vaccine and the MVA/HIV62B vaccine in healthy, HIV-1-uninfected adults who previously received MVA/HIV62B in DNA/MVA or MVA/MVA vaccine regimens as part of the HVTN 205 study.

Participants in this study will be assigned to one of five groups based on their previous vaccine regimen received in HVTN 205. Depending on their group, participants will receive the MVA/HIV62B vaccine, the AIDSVAX B/E vaccine, or both the MVA/HIV62B vaccine and the AIDSVAX B/E vaccine. All participants will receive their assigned vaccines at study entry (Day 0) and Month 4. Participants will attend several study visits through Month 10. Visits will include physical examinations, blood collection, HIV testing and risk reduction counseling, and interviews and questionnaires. Optional procedures at some visits include collection of rectal fluids, cervical fluids, and semen. Study staff will contact participants 2 years following the initial study injection for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria:

* Age of 18 to 55 years
* Prior participation in HVTN 205 with assignment to treatment (not placebo) arm:

  1. Assigned to HVTN 205 Group 1 or Group 3, and received all 4 scheduled vaccinations (2 injections of pGA2/JS7 DNA (months 0, 2) and 2 injections of MVA/HIV62 (months 4, 6); OR
  2. Assigned to HVTN 205 Group 4, and received at least vaccinations 1, 2 and 4 (3 injections of MVA/HIV62 at months 0, 2 and 6).
* Access to a participating HVTN clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted 2 years following initial study injection.
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

Laboratory Inclusion Values:

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.
* Cardiac Troponin T or I (cTnT or cTnI) does not exceed the institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: Participants must have a negative test result for HIV infection following the HVTN Lab Program's in-study HIV testing algorithm, prior to initial enrollment.
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus Ab (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (more information is available in the protocol) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Any other contraceptive method approved by the HVTN 114 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40
* Volunteer has 2 or more of the following cardiac risk factors:

  * Participant report of history of elevated blood cholesterol defined as fasting LDL greater than 160 mg/dL;
  * First degree relative (eg, mother, father, brother, or sister) who had coronary artery disease before the age of 50 years;
  * Current smoker; or
  * BMI greater than or equal to 35
* Pregnant or breastfeeding
* Active duty and reserve U.S. military personnel

Vaccines and Other Injections

* Any clinically significant AE related to vaccination in HVTN 205, for which revaccination would be a safety concern such as any grade 3 or 4 related AE
* Smallpox vaccine received within the last 5 years
* HIV vaccine(s) received in a prior HIV vaccine trial other than HVTN 205. For HVTN 205 participants who have subsequently received control/placebo in another HIV vaccine trial, the HVTN 114 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 114 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 114 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Hypersensitivity to eggs or egg products
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease (eg, myositis)
* Immunodeficiency

Cardiac

* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
* ECG with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, as determined by a contract ECG Lab or cardiologist, including any of the following: (1) conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS greater than or equal to 120 ms, PR interval greater than or equal to 220ms, any 2nd or 3rd degree AV block, or QTc prolongation (greater than 450ms)); (2) repolarization (ST segment or T wave) abnormality that will interfere with the assessment of myo/pericarditis; (3) significant atrial or ventricular arrhythmia; (4) frequent atrial or ventricular ectopy (eg, frequent premature atrial contractions, 2 premature ventricular contractions in a row); (5) ST elevation consistent with ischemia; (6) evidence of past or evolving myocardial infarction

Clinically Significant Medical Conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

  * Exclude a volunteer who:
  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goepfert, Study Chair — University of Alabama at Birmingham
Locations (9):
- United States (7):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Peru (2):
  - ACSA CRS, Iquitos, Maynas
  - Barranco CRS, Lima

REFERENCES:
- [Background] Huang Y, Seaton KE, Casapia M, Polakowski L, De Rosa SC, Cohen K, Yu C, Elizaga M, Paez C, Miner MD, Kelley CF, Maenza J, Keefer M, Lama JR, Sobieszczyk M, Buchbinder S, Baden LR, Lee C, Gulati V, Sinangil F, Montefiori D, McElrath MJ, Tomaras GD, Robinson HL, Goepfert P; NIAID-funded HIV Vaccine Trials Network (HVTN) 114 Study Team. AIDSVAX protein boost improves breadth and magnitude of vaccine-induced HIV-1 envelope-specific responses after a 7-year rest period. Vaccine. 2021 Jul 30;39(33):4641-4650. doi: 10.1016/j.vaccine.2021.06.066. Epub 2021 Jul 3. PMID 34229888
- [Derived] Fischinger S, Cizmeci D, Deng D, Grant SP, Frahm N, McElrath J, Fuchs J, Bart PA, Pantaleo G, Keefer M, O Hahn W, Rouphael N, Churchyard G, Moodie Z, Donastorg Y, Streeck H, Alter G. Sequence and vector shapes vaccine induced antibody effector functions in HIV vaccine trials. PLoS Pathog. 2021 Nov 29;17(11):e1010016. doi: 10.1371/journal.ppat.1010016. eCollection 2021 Nov. PMID 34843602

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Boost: MVA/HIV62B mo(0,4) post HVTN 205 MMM
- Group 2: Boost: MVA/HIV62B + AIDSVAX B/E mo(0,4) post HVTN 205 MMM
- Group 3: Boost: MVA/HIV62B mo(0,4) post HVTN 205 DDMM
- Group 4: Boost: MVA/HIV62B + AIDSVAX B/E mo(0,4) post HVTN 205 DDMM
- Group 5: Boost: AIDSVAX B/E mo(0,4) post HVTN 205 DDMM
Period: Overall Study
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Started | 4 | 4 | 6 | 6 | 7
Month 0.5 | 3 | 4 | 6 | 6 | 7
Month 4.5 | 3 | 4 | 6 | 6 | 7
Month 10 | 3 | 3 | 6 | 5 | 7
Completed | 3 | 4 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Total
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 27
Age, Continuous [Median (Full Range); unit: years] | 32 [29 to 37] | 32 [26 to 35] | 32 [27 to 39] | 30 [26 to 54] | 36 [25 to 43] | 33 [25 to 54]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 | 0 | 0 | 0 | 0 | 0 | 0
  21 - 30 | 2 | 2 | 1 | 3 | 2 | 10
  31 - 40 | 2 | 2 | 5 | 2 | 3 | 14
  41 - 50 | 0 | 0 | 0 | 0 | 2 | 2
  Over 50 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 3 | 4 | 16
  Male | 2 | 1 | 2 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 4 | 4 | 11
  Not Hispanic or Latino | 4 | 4 | 3 | 2 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 1 | 3
  White | 2 | 3 | 2 | 3 | 2 | 12
  More than one race | 0 | 1 | 3 | 3 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 3 | 3 | 3 | 17
  Peru | 0 | 0 | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms of the Left Arm (MVA/HIV62B or Placebo)
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 [November 2014], The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after the boost at Month 0 and Month 4
Population: The "overall number of participants analyzed" represents participants enrolled and received MVA/HIV62B or placebo. However, one participant in T5 received MVA/HIV62B placebo in the right arm. Hence no left arm reactogenicity data was collected for the participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6
Participants
  Pain: None | 0 | 0 | 0 | 0 | 2
  Pain: Mild | 1 | 0 | 3 | 5 | 4
  Pain: Moderate | 3 | 4 | 3 | 1 | 0
  Pain: Severe | 0 | 0 | 0 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Tenderness: None | 0 | 0 | 0 | 1 | 4
  Tenderness: Mild | 3 | 2 | 3 | 4 | 1
  Tenderness: Moderate | 1 | 2 | 3 | 1 | 1
  Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 0 | 0 | 0 | 0 | 2
  Pain and/or Tenderness: Mild | 1 | 0 | 3 | 5 | 3
  Pain and/or Tenderness: Moderate | 3 | 4 | 3 | 1 | 1
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema: None | 4 | 4 | 3 | 6 | 6
  Erythema: Mild | 0 | 0 | 1 | 0 | 0
  Erythema: Moderate | 0 | 0 | 1 | 0 | 0
  Erythema: Severe | 0 | 0 | 1 | 0 | 0
  Erythema: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Induration: None | 4 | 4 | 3 | 6 | 5
  Induration: Mild | 0 | 0 | 1 | 0 | 1
  Induration: Moderate | 0 | 0 | 2 | 0 | 0
  Induration: Severe | 0 | 0 | 0 | 0 | 0
  Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 4 | 4 | 3 | 6 | 5
  Erythema and/or Induration: Mild | 0 | 0 | 1 | 0 | 1
  Erythema and/or Induration: Moderate | 0 | 0 | 1 | 0 | 0
  Erythema and/or Induration: Severe | 0 | 0 | 1 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms of the Right Arm (AIDSVAX B/E or Placebo)
Description: as for outcome 1
Time Frame: Measured through 3 days after the boost at Month 0 and Month 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7
Participants
  Pain: None | 3 | 0 | 4 | 2 | 1
  Pain: Mild | 0 | 4 | 2 | 4 | 5
  Pain: Moderate | 1 | 0 | 0 | 0 | 1
  Pain: Severe | 0 | 0 | 0 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Tenderness: None | 3 | 0 | 5 | 3 | 1
  Tenderness: Mild | 1 | 2 | 1 | 2 | 4
  Tenderness: Moderate | 0 | 2 | 0 | 1 | 2
  Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 3 | 0 | 4 | 1 | 1
  Pain and/or Tenderness: Mild | 0 | 2 | 2 | 4 | 4
  Pain and/or Tenderness: Moderate | 1 | 2 | 0 | 1 | 2
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema: None | 4 | 4 | 6 | 6 | 7
  Erythema: Mild | 0 | 0 | 0 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0 | 0 | 0
  Erythema: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Induration: None | 4 | 4 | 6 | 6 | 6
  Induration: Mild | 0 | 0 | 0 | 0 | 1
  Induration: Moderate | 0 | 0 | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0 | 0 | 0
  Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 4 | 4 | 6 | 6 | 6
  Erythema and/or Induration: Mild | 0 | 0 | 0 | 0 | 1
  Erythema and/or Induration: Moderate | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms During the Boost Regimen
Description: as for outcome 1
Time Frame: Measured through Month Measured through 3 days after each boost at Month 0 and 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7
Participants
  Malaise and/or fatigue: None | 1 | 0 | 2 | 2 | 6
  Malaise and/or fatigue: Mild | 1 | 2 | 1 | 2 | 0
  Malaise and/or fatigue: Moderate | 2 | 2 | 3 | 1 | 1
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 1 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 1 | 1 | 2 | 2 | 5
  Myalgia: Mild | 0 | 1 | 0 | 1 | 2
  Myalgia: Moderate | 3 | 2 | 4 | 2 | 0
  Myalgia: Severe | 0 | 0 | 0 | 1 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Headache: None | 1 | 2 | 2 | 2 | 7
  Headache: Mild | 2 | 1 | 1 | 2 | 0
  Headache: Moderate | 1 | 1 | 3 | 1 | 0
  Headache: Severe | 0 | 0 | 0 | 1 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Nausea: None | 3 | 2 | 6 | 5 | 7
  Nausea: Mild | 1 | 2 | 0 | 1 | 0
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Vomiting: None | 4 | 4 | 6 | 6 | 7
  Vomiting: Mild | 0 | 0 | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Chills: None | 2 | 0 | 3 | 1 | 6
  Chills: Mild | 1 | 3 | 0 | 2 | 0
  Chills: Moderate | 1 | 1 | 3 | 2 | 1
  Chills: Severe | 0 | 0 | 0 | 1 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 2 | 0 | 4 | 4 | 6
  Arthralgia: Mild | 0 | 2 | 1 | 1 | 1
  Arthralgia: Moderate | 2 | 2 | 1 | 1 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 0 | 0 | 1 | 1 | 4
  Max. Systemic Symptoms: Mild | 1 | 2 | 1 | 1 | 1
  Max. Systemic Symptoms: Moderate | 3 | 2 | 4 | 3 | 2
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 1 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 3 | 3 | 4 | 6
  Temperature: Mild | 1 | 0 | 2 | 0 | 1
  Temperature: Moderate | 0 | 0 | 1 | 2 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: From the study termination form, early termination reasons associated with an AE or reactogenicity are tabulated by treatment arm
Time Frame: Measured through Month 10
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7
Participants
  Adverse event or reactogenicity | 0 | 0 | 0 | 0 | 0
  No adverse event or reactogenicity | 0 | 0 | 0 | 0 | 0
  Do not know | 1 | 0 | 0 | 0 | 0
  No termination | 3 | 4 | 6 | 6 | 7

5. Primary Outcome: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm
Time Frame: Measured through the Month 4 boost
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7
Participants
  Clinical Event | 0 | 0 | 0 | 0 | 0
  Reactogenicity | 0 | 1 | 0 | 0 | 0
  Other reason | 1 | 0 | 0 | 0 | 0
  No discontinuation | 3 | 3 | 6 | 6 | 7

6. Primary Outcome: Chemistry and Hematology Laboratory Measures, for Each Boost: Alkaline Phosphatase, AST, ALT in U/L
Description: For each chemistry laboratory measure, summary statistics were presented by analyte and treatment group for the overall population.
Time Frame: Measured during screening, and 2 weeks after each boost at Month 0 and 4
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7
U/L
  Alkaline Phosphatase (U/L)- Screening | 54.5 [50.5 to 61] | 63.5 [48.5 to 66.5] | 91 [52 to 99] | 78.5 [45 to 99] | 55 [39 to 112]
  Alkaline Phosphatase (U/L)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Alkaline Phosphatase (U/L)- Day14 | 59 [56 to 59] | 68.5 [49.5 to 74.5] | 73 [58 to 101] | 57 [40 to 83] | 52 [38 to 105]
  Alkaline Phosphatase (U/L)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Alkaline Phosphatase (U/L)- Day126 | 58 [55 to 69] | 63 [45.5 to 77] | 69 [64 to 73] | 72 [40 to 84] | 53 [38 to 73]
  AST (U/L)- Screening | 16.5 [12.5 to 21.5] | 16.5 [14 to 20] | 20 [17 to 30] | 17.5 [15 to 20] | 24 [20 to 25]
  AST (U/L)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  AST (U/L)- Day14 | 18 [14 to 28] | 15.5 [13.5 to 21] | 26 [18 to 27] | 21 [18 to 22] | 24 [18 to 30]
  AST (U/L)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  AST (U/L)- Day126 | 18 [13 to 25] | 19 [16.5 to 21.5] | 17 [15 to 25] | 22.5 [20 to 26] | 22 [18 to 28]
  ALT (SGPT) (U/L)- Screening | 15.5 [11.5 to 22.5] | 16.5 [13.5 to 20] | 23 [14 to 32] | 14.5 [13 to 23] | 26 [15 to 32]
  ALT (SGPT) (U/L)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  ALT (SGPT) (U/L)- Day14 | 18 [10 to 20] | 16 [12.5 to 19.5] | 23 [16 to 29] | 21.5 [16 to 25] | 23 [13 to 34]
  ALT (SGPT) (U/L)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  ALT (SGPT) (U/L)- Day126 | 14 [9 to 16] | 15.5 [14.5 to 23.5] | 16.5 [16 to 29] | 22.5 [15 to 37] | 28 [15 to 37]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures, for Each Boost: Hemoglobin, Creatinine in g/dL
Description: as for outcome 6
Time Frame: Measured during screening, and 2 weeks after each boost at Month 0 and 4
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7
g/dL
  Hemoglobin (g/dL)- Screening | 14 [12.75 to 14.95] | 13.6 [12.95 to 14.05] | 13 [12.3 to 15.8] | 14.5 [13.8 to 15.1] | 14 [12.2 to 15.1]
  Hemoglobin (g/dL)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Hemoglobin (g/dL)- Day14 | 15 [11.4 to 15.6] | 13.55 [13.15 to 14.05] | 12.85 [12.5 to 14.6] | 14.05 [13 to 14.9] | 12.9 [12.1 to 14.7]
  Hemoglobin (g/dL)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Hemoglobin (g/dL)- Day126 | 14.9 [11.3 to 15.8] | 13.9 [13.65 to 14.15] | 13.2 [12.2 to 14.5] | 14.65 [13.7 to 14.8] | 12.8 [12.2 to 14.3]
  Creatinine (g/dL)- Screening | 0.000785 [0.00075 to 0.00085] | 0.000805 [0.000715 to 0.000845] | 0.00072 [0.00071 to 0.0009] | 0.000755 [0.00063 to 0.00088] | 0.00085 [0.00055 to 0.00091]
  Creatinine (g/dL)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Creatinine (g/dL)- Day14 | 0.0008 [0.00068 to 0.0008] | 0.000795 [0.000765 to 0.000865] | 0.0008 [0.00072 to 0.00099] | 0.000835 [0.00053 to 0.00093] | 0.00092 [0.00063 to 0.00096]
  Creatinine (g/dL)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Creatinine (g/dL)- Day126 | 0.0009 [0.00077 to 0.00094] | 0.00075 [0.000715 to 0.00079] | 0.000725 [0.00064 to 0.0009] | 0.000785 [0.0006 to 0.00091] | 0.00085 [0.0006 to 0.0009]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures, for Each Boost: WBC, Platelets, Lymphocytes, Neutrophils
Description: as for outcome 6
Time Frame: Measured during screening, and 2 weeks after each boost at Month 0 and 4
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7
thousand cells/cubic mm
  WBC (1000/cubic mm)- Screening | 5.8 [5.45 to 7.23] | 6.27 [4.115 to 8.65] | 6.875 [5.87 to 8] | 6.4 [5.5 to 7.1] | 5.8 [4.84 to 8.7]
  WBC (1000/cubic mm)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  WBC (1000/cubic mm)- Day14 | 6.3 [4.3 to 9.97] | 6.5 [4.745 to 9.225] | 7.555 [5.91 to 8.9] | 5.65 [4.7 to 8.4] | 7.4 [4.27 to 7.98]
  WBC (1000/cubic mm)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  WBC (1000/cubic mm)- Day126 | 7 [4.4 to 10.65] | 7.47 [4.56 to 9.875] | 7.25 [5.55 to 9.62] | 4.85 [4.2 to 6] | 5.6 [4.47 to 8.1]
  Platelets (1000/cubic mm)- Screening | 220.8 [195 to 239.3] | 256.5 [216.5 to 287.5] | 329.85 [295 to 368] | 269.5 [247 to 296] | 266 [191 to 320]
  Platelets (1000/cubic mm)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Platelets (1000/cubic mm)- Day14 | 251 [152 to 252.2] | 309.5 [253 to 383.5] | 325.6 [308 to 338] | 306 [271 to 321] | 267 [211 to 340]
  Platelets (1000/cubic mm)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Platelets (1000/cubic mm)- Day126 | 234.5 [179 to 244] | 259 [229.5 to 347] | 340 [314 to 359] | 279 [254 to 296] | 285 [228 to 373]
  Lymphocytes (cells/cubic mm)- Screening | 1423.5 [1144 to 2256] | 2426 [1785 to 3111] | 2042 [1420 to 2400] | 2055.5 [1557 to 2268] | 1950 [1566 to 2262]
  Lymphocytes (cells/cubic mm)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Lymphocytes (cells/cubic mm)- Day14 | 1449 [920 to 2991] | 2483.5 [1825 to 2913.5] | 2153.5 [1980 to 2300] | 1798 [1512 to 2268] | 2075 [1779 to 2220]
  Lymphocytes (cells/cubic mm)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Lymphocytes (cells/cubic mm)- Day126 | 1855 [1580 to 3089] | 2670 [1770 to 2922] | 2084 [1891 to 2688] | 1800 [1617 to 2129] | 1652 [1370 to 2592]
  Neutrophils (cells/cubic mm)- Screening | 4151.5 [3545 to 4694] | 3260 [1777 to 4740] | 4195 [3690 to 4960] | 3803 [2806 to 4261] | 3229 [2770 to 4823]
  Neutrophils (cells/cubic mm)- Day14: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Neutrophils (cells/cubic mm)- Day14 | 4190 [2636 to 6281] | 3855 [2076 to 5785] | 4759.5 [3290 to 4895] | 3587.5 [2820 to 4704] | 4187 [2390 to 4944]
  Neutrophils (cells/cubic mm)- Day126: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7
  Neutrophils (cells/cubic mm)- Day126 | 4473 [2204 to 6710] | 4162.5 [2037.5 to 6545] | 4254.5 [3320 to 5800] | 2364 [2201 to 3720] | 3584 [2590 to 4455]

9. Primary Outcome: Occurrence of Env-specific IgG Responses for gp120, gp41, V1/V2, and the IDR of gp41 at 2 Weeks After Each Boost
Description: Serum HIV-1-specific IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation. The responses to the IDR of gp41 was not assayed.
Time Frame: Measured at Month 0.5 and 4.5
Population: "Overall Number of Participants Analyzed" includes the HIV uninfected participants with samples collected at the months 0.5 or 4.5 immunogenicity timepoint. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Group 6: Boost: MVA/HIV62B at mo(0,4)
- Group 7: Boost: MVA/HIV62B + AIDSVAX B/E at mo(0,4)
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Participants
  Con 6 gp120/B at Month 0.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con 6 gp120/B at Month 0.5 | 1 | 3 | 2 | 4 | 7 | 3 | 7
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con 6 gp120/B at Month 4.5 | 0 | 3 | 2 | 4 | 7 | 2 | 7
  Con S gp140 CFI at Month 0.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con S gp140 CFI at Month 0.5 | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con S gp140 CFI at Month 4.5 | 2 | 3 | 4 | 4 | 7 | 6 | 7
  gp41 at Month 0.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  gp41 at Month 0.5 | 2 | 3 | 4 | 4 | 1 | 6 | 7
  gp41 at Month 4.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  gp41 at Month 4.5 | 2 | 3 | 4 | 4 | 1 | 6 | 7
  gp70_B.CaseA_V1_V2 at Month 0.5: number analyzed (Participants) | 2 | 3 | 5 | 6 | 7 | 7 | 9
  gp70_B.CaseA_V1_V2 at Month 0.5 | 1 | 1 | 0 | 4 | 4 | 1 | 5
  gp70_B.CaseA_V1_V2 at Month 4.5: number analyzed (Participants) | 2 | 3 | 5 | 6 | 7 | 7 | 9
  gp70_B.CaseA_V1_V2 at Month 4.5 | 2 | 2 | 0 | 6 | 6 | 2 | 8

10. Primary Outcome: Level of Env-specific IgG Responses for gp120, gp41, V1/V2, and the IDR of gp41 at 2 Weeks After Each Boost
Description: as for outcome 9
Time Frame: Measured at Month 0.5 and 4.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
fluorescence unit relative to background
  Con 6 gp120/B at Month 0.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con 6 gp120/B at Month 0.5 | 220.875 [1 to 440.75] | 8614 [5879 to 26686.25] | 196 [74.75 to 244.75] | 28087 [26883.5 to 29222.25] | 23785.75 [5630.25 to 27778.5] | 196 [1 to 246] | 26686.25 [8614 to 28563.75]
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con 6 gp120/B at Month 4.5 | 83.25 [41.5 to 125] | 5747.5 [2239 to 22439] | 172 [112.875 to 288] | 24074.75 [22735.25 to 27543.625] | 18736.75 [15876.75 to 27143.75] | 139 [72.75 to 191] | 22439 [5747.5 to 24689.75]
  Con S gp140 CFI at Month 0.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con S gp140 CFI at Month 0.5 | 17731.875 [4716.5 to 30747.25] | 32346.75 [29849 to 32654.25] | 14689.25 [10853.125 to 17512.5] | 31583.375 [31444.875 to 32142.75] | 30936.5 [27708.25 to 31563.5] | 14689.25 [8404 to 18948.75] | 31707.5 [31430.5 to 32578]
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  Con S gp140 CFI at Month 4.5 | 14087.75 [7946.25 to 20229.25] | 25825.5 [25002.5 to 32600.25] | 23503.125 [15374.375 to 25633.75] | 30404.5 [29352.5 to 31714.75] | 28886.5 [21889 to 30798.25] | 21358.125 [8261.75 to 24519.25] | 29998.5 [25825.5 to 32600.25]
  gp41 at Month 0.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  gp41 at Month 0.5 | 19616.625 [6577.75 to 32655.5] | 32345 [29809 to 32647.25] | 17144.25 [9655.625 to 26767.375] | 27552.75 [15555.375 to 30144.875] | 2412.5 [296.75 to 7347] | 17144.25 [8024.5 to 30533] | 29809 [27392.5 to 32576.75]
  gp41 at Month 4.5: number analyzed (Participants) | 2 | 3 | 4 | 4 | 7 | 6 | 7
  gp41 at Month 4.5 | 18819.125 [10370.5 to 27267.75] | 31713 [28452.25 to 32588.5] | 24536.5 [12926.25 to 29876.375] | 27619.125 [25238.5 to 29852.625] | 2084.25 [245 to 5110] | 23852.25 [10370.5 to 28636.25] | 28452.25 [27056.75 to 31713]
  gp70_B.CaseA_V1_V2 at Month 0.5: number analyzed (Participants) | 2 | 3 | 5 | 6 | 7 | 7 | 9
  gp70_B.CaseA_V1_V2 at Month 0.5 | 565.125 [15 to 1115.25] | 87.25 [1 to 1985.75] | 1 [1 to 1] | 1045.875 [23.25 to 26299] | 181.75 [1 to 4502] | 1 [1 to 15] | 611.75 [23.25 to 1985.75]
  gp70_B.CaseA_V1_V2 at Month 4.5: number analyzed (Participants) | 2 | 3 | 5 | 6 | 7 | 7 | 9
  gp70_B.CaseA_V1_V2 at Month 4.5 | 605.5 [332.25 to 878.75] | 15735 [1 to 23942.5] | 1 [1 to 3.25] | 4909 [3774.75 to 10989.75] | 11250.75 [2338.75 to 25894.5] | 3.25 [1 to 332.25] | 4948.75 [3774.75 to 15735]

11. Primary Outcome: Occurrence of Env-specific IgG3 Responses for gp120, gp41, V1/V2, and the IDR of gp41 at 2 Weeks After Each Boost
Description: Serum HIV-1-specific IgG3 responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation. The responses to the IDR of gp41 was not assayed.
Time Frame: Measured at Month 0.5 and 4.5
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Participants
  Con 6 gp120/B at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con 6 gp120/B at Month 0.5 | 0 | 0 | 0 | 2 | 2 | 0 | 2
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con 6 gp120/B at Month 4.5 | 0 | 1 | 0 | 2 | 2 | 0 | 3
  Con S gp140 CFI at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con S gp140 CFI at Month 0.5 | 2 | 3 | 4 | 4 | 2 | 6 | 7
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con S gp140 CFI at Month 4.5 | 2 | 2 | 4 | 4 | 1 | 6 | 6
  gp41 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp41 at Month 0.5 | 2 | 4 | 3 | 5 | 0 | 5 | 9
  gp41 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp41 at Month 4.5 | 2 | 2 | 4 | 5 | 0 | 6 | 7
  gp70_B.CaseA_V1_V2 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp70_B.CaseA_V1_V2 at Month 0.5 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  gp70_B.CaseA_V1_V2 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp70_B.CaseA_V1_V2 at Month 4.5 | 0 | 2 | 0 | 4 | 1 | 0 | 6

12. Primary Outcome: Level of Env-specific IgG3 Responses for gp120, gp41, V1/V2, and the IDR of gp41 at 2 Weeks After Each Boost
Description: as for outcome 11
Time Frame: Measured at Month 0.5 and 4.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
fluorescence unit relative to background
  Con 6 gp120/B at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con 6 gp120/B at Month 0.5 | 1 [1 to 1] | 5.875 [3.375 to 11.375] | 1 [1 to 1] | 8 [4.25 to 126.75] | 6 [3 to 370.25] | 1 [1 to 1] | 5.875 [4.25 to 16.5]
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con 6 gp120/B at Month 4.5 | 1 [1 to 1] | 2.75 [1 to 394.25] | 1 [1 to 1] | 55.125 [20.75 to 165] | 26.25 [12.5 to 106.25] | 1 [1 to 1] | 31.375 [1 to 165]
  Con S gp140 CFI at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con S gp140 CFI at Month 0.5 | 113.75 [43 to 6460.5] | 236.125 [134.875 to 1394.25] | 218.375 [42.5 to 647.25] | 705.75 [81.5 to 6505.5] | 26 [14 to 444] | 129.25 [43 to 647.25] | 236.125 [81.5 to 2541.75]
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Con S gp140 CFI at Month 4.5 | 162.25 [47.25 to 1909.25] | 230.125 [14.125 to 1464.125] | 279.5 [45.75 to 636.5] | 558.5 [93.5 to 3852.25] | 17.5 [12 to 56] | 162.25 [47.25 to 636.5] | 473.875 [37.75 to 2487]
  gp41 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp41 at Month 0.5 | 4137.5 [234.25 to 15416.5] | 870.75 [701.625 to 5744.125] | 525.875 [100.5 to 12995.25] | 794.375 [513 to 1269.75] | 41 [23 to 56.5] | 889 [162.75 to 12995.25] | 845.25 [619.5 to 1269.75]
  gp41 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp41 at Month 4.5 | 1338.25 [181.25 to 4636.75] | 770.5 [211.875 to 3107.5] | 1770.5 [142.5 to 7997.5] | 1942.25 [309.75 to 17175.5] | 29 [21.25 to 59] | 1343.75 [181.25 to 4636.75] | 803.5 [258.75 to 4932.75]
  gp70_B.CaseA_V1_V2 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp70_B.CaseA_V1_V2 at Month 0.5 | 1 [1 to 1] | 32.5 [1 to 224.625] | 1 [1 to 1] | 1 [1 to 57] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 64]
  gp70_B.CaseA_V1_V2 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  gp70_B.CaseA_V1_V2 at Month 4.5 | 1 [1 to 1] | 92.875 [22 to 3889.125] | 1 [1 to 1] | 113.125 [15.25 to 162] | 9.75 [1 to 25.25] | 1 [1 to 1] | 113.125 [15.25 to 162]

13. Primary Outcome: Occurrence of Env-specific IgA Responses for gp120, gp41, V1V2, and the IDR of gp41 at 2 Weeks After Each Boost
Description: Serum HIV-1-specific IgA responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation. IgA responses to V1V2 and the IDR of gp41 were not assayed.
Time Frame: Measured at Month 0.5 and 4.5
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Participants
  Con 6 gp120/B at Month 0.5: number analyzed (Participants) | 2 | 4 | 5 | 6 | 7 | 7 | 10
  Con 6 gp120/B at Month 0.5 | 0 | 3 | 0 | 4 | 6 | 0 | 7
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 2 | 4 | 5 | 5 | 6 | 7 | 9
  Con 6 gp120/B at Month 4.5 | 0 | 1 | 0 | 4 | 3 | 0 | 5
  Con S gp140 CFI at Month 0.5: number analyzed (Participants) | 2 | 4 | 5 | 6 | 7 | 7 | 10
  Con S gp140 CFI at Month 0.5 | 1 | 3 | 0 | 5 | 7 | 1 | 8
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 2 | 4 | 5 | 5 | 6 | 7 | 9
  Con S gp140 CFI at Month 4.5 | 1 | 1 | 0 | 5 | 4 | 1 | 6
  gp41 at Month 0.5: number analyzed (Participants) | 2 | 4 | 5 | 6 | 7 | 7 | 10
  gp41 at Month 0.5 | 1 | 1 | 0 | 2 | 2 | 1 | 3
  gp41 at Month 4.5: number analyzed (Participants) | 2 | 4 | 5 | 5 | 6 | 7 | 9
  gp41 at Month 4.5 | 0 | 2 | 0 | 2 | 0 | 0 | 4

14. Primary Outcome: Level of Env-specific IgA Responses for gp120, gp41, V1V2, and the IDR of gp41 at 2 Weeks After Each Boost
Description: as for outcome 13
Time Frame: Measured at Month 0.5 and 4.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
fluorescence unit relative to background
  Con 6 gp120/B at Month 0.5: number analyzed (Participants) | 2 | 4 | 5 | 6 | 7 | 7 | 10
  Con 6 gp120/B at Month 0.5 | 1 [1 to 1] | 3035.25 [110.625 to 12698.75] | 1 [1 to 1] | 4259.75 [608.25 to 13610.5] | 808.25 [263.75 to 5132.5] | 1 [1 to 1] | 4136.375 [220.25 to 13610.5]
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 2 | 4 | 5 | 5 | 6 | 7 | 9
  Con 6 gp120/B at Month 4.5 | 1 [1 to 1] | 35.75 [1 to 3582.125] | 1 [1 to 1] | 482.25 [241.5 to 837.25] | 571.75 [14.25 to 2904] | 1 [1 to 1] | 241.5 [70.5 to 837.25]
  Con S gp140 CFI at Month 0.5: number analyzed (Participants) | 2 | 4 | 5 | 6 | 7 | 7 | 10
  Con S gp140 CFI at Month 0.5 | 162.5 [1 to 324] | 12600.125 [196.875 to 26081.25] | 1 [1 to 1] | 12951.625 [139.75 to 23511] | 1577.25 [1095 to 19696.25] | 1 [1 to 2.75] | 12951.625 [139.75 to 24807.5]
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 2 | 4 | 5 | 5 | 6 | 7 | 9
  Con S gp140 CFI at Month 4.5 | 161.375 [1 to 321.75] | 3.625 [1 to 4473] | 1 [1 to 1] | 554.75 [304.75 to 750.25] | 711.5 [94.25 to 2831.25] | 1 [1 to 6.25] | 304.75 [6.25 to 750.25]
  gp41 at Month 0.5: number analyzed (Participants) | 2 | 4 | 5 | 6 | 7 | 7 | 10
  gp41 at Month 0.5 | 235.5 [1 to 470] | 362.5 [80.625 to 708.125] | 72.75 [22.5 to 127.25] | 484.875 [101.75 to 1094] | 39.25 [1 to 212.5] | 72.75 [1 to 228.25] | 431.875 [101.75 to 851.5]
  gp41 at Month 4.5: number analyzed (Participants) | 2 | 4 | 5 | 5 | 6 | 7 | 9
  gp41 at Month 4.5 | 193.125 [1 to 385.25] | 119.375 [1 to 288.625] | 30.5 [26 to 37.5] | 206.75 [98.25 to 277.75] | 46.375 [1 to 185.5] | 30.5 [1 to 131] | 206.75 [1 to 277.75]

15. Primary Outcome: Occurrence of Neutralizing Ab Titers and Breadth Against the Env Vaccine Strain and Heterologous Tier 1 Strains at 2 Weeks After Each Boost
Description: Neutralizing antibodies against HIV-1 were measured as a function of reductions in Tat-regulated luciferase (Luc) reporter gene expression in TZM-bl cells. The assay measured neutralization titers against a panel of autologous and heterologous Env-pseudotyped viruses.
Time Frame: Measured at Month 0.5 and 4.5
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Participants
  ADA at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  ADA at Month 0.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  ADA at Month 4.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CM244.c01 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  CM244.c01 at Month 0.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CM244.c01 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  CM244.c01 at Month 4.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MN.3 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  MN.3 at Month 0.5 | 2 | 4 | 2 | 6 | 7 | 4 | 10
  MN.3 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  MN.3 at Month 4.5 | 1 | 3 | 3 | 6 | 7 | 4 | 9
  TH023.6 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  TH023.6 at Month 0.5 | 0 | 1 | 0 | 4 | 2 | 0 | 5
  TH023.6 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  TH023.6 at Month 4.5 | 0 | 2 | 0 | 3 | 4 | 0 | 5

16. Primary Outcome: Level of Neutralizing Ab Titers and Breadth Against the Env Vaccine Strain and Heterologous Tier 1 Strains at 2 Weeks After Each Boost
Description: Neutralizing antibodies against HIV-1 were measured as a function of reductions in Tat-regulated luciferase (Luc) reporter gene expression in TZM-bl cells. The assay measured neutralization titers against a panel of autologous and heterologous Env-pseudotyped viruses. A serum neutralization titer was defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% (ID50) relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). Titer < 10 is truncated at 5.
Time Frame: Measured at Month 0.5 and 4.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Dilution factor
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Dilution factor
  ADA at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  ADA at Month 0.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  ADA at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  ADA at Month 4.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CM244.c01 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  CM244.c01 at Month 0.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CM244.c01 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  CM244.c01 at Month 4.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  MN.3 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  MN.3 at Month 0.5 | 37 [5 to 60] | 1388.5 [482.5 to 12007] | 7.5 [5 to 16] | 11414.5 [6171 to 21870] | 6608 [635 to 14666] | 10 [5 to 37] | 7485 [1716 to 21870]
  MN.3 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  MN.3 at Month 4.5 | 5 [5 to 50] | 196 [53 to 625.5] | 8.5 [5 to 28] | 944.5 [499 to 1666] | 996 [138 to 1285] | 5 [5 to 28] | 522.5 [291 to 1343]
  TH023.6 at Month 0.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  TH023.6 at Month 0.5 | 5 [5 to 5] | 5 [5 to 11] | 5 [5 to 5] | 18 [5 to 24] | 5 [5 to 11] | 5 [5 to 5] | 8.5 [5 to 24]
  TH023.6 at Month 4.5: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  TH023.6 at Month 4.5 | 5 [5 to 5] | 80 [5 to 156.5] | 5 [5 to 5] | 16 [5 to 41] | 23 [5 to 145] | 5 [5 to 5] | 16 [5 to 98]

17. Secondary Outcome: Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine 2 Weeks After Each Boost
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers after peptide stimulation minus % cells expressing markers after no stimulation. Response positivity is derived by testing if the number of cells expressing the marker is equal in the stimulated vs. unstimulated cells. Response is positive if the one-sided Fisher's exact test (discrete Bonferroni adjustment over the peptide pools) p<=0.00001. The Fisher's exact test is not applied to compare between endpoints. Data are excluded if the blood draw date was outside the visit window, the participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high. The responses at month 0.5 was not assayed.
Time Frame: Measured at Month 4.5
Population: "Overall Number of Participants Analyzed" includes the HIV uninfected participants with samples collected at the month 4.5 immunogenicity timepoint. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Participants
  Any Env PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Any Env PTEg | 0 | 2 | 2 | 5 | 4 | 2 | 7
  Any Gag PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Any Gag PTEg | 2 | 2 | 6 | 5 | 1 | 8 | 7
  Any PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Any PTEg | 2 | 2 | 6 | 5 | 4 | 8 | 7
  Env-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Env-1-PTEg | 0 | 2 | 2 | 5 | 3 | 2 | 7
  Env-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Env-2-PTEg | 0 | 0 | 1 | 3 | 3 | 1 | 3
  Env-3-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Env-3-PTEg | 0 | 1 | 0 | 3 | 1 | 0 | 4
  Gag-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Gag-1-PTEg | 2 | 2 | 6 | 5 | 1 | 8 | 7
  Gag-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Gag-2-PTEg | 0 | 0 | 3 | 4 | 0 | 3 | 4

18. Secondary Outcome: Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine 2 Weeks After Each Boost
Description: as for outcome 17
Time Frame: Measured at Month 4.5
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
% CD4+ T-cells
  Any Env PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Any Env PTEg | 0.032 [0.014 to 0.033] | 0.074 [0.05 to 0.082] | 0.048 [0.04 to 0.131] | 0.142 [0.058 to 0.218] | 0.083 [0.036 to 0.12] | 0.04 [0.033 to 0.05] | 0.082 [0.058 to 0.165]
  Any Gag PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Any Gag PTEg | 0.06 [0.04 to 0.108] | 0.054 [0.035 to 0.062] | 0.163 [0.101 to 0.185] | 0.196 [0.053 to 0.272] | 0.015 [0 to 0.031] | 0.108 [0.06 to 0.165] | 0.062 [0.048 to 0.211]
  Any PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Any PTEg | 0.074 [0.072 to 0.142] | 0.129 [0.091 to 0.138] | 0.218 [0.141 to 0.325] | 0.338 [0.111 to 0.509] | 0.085 [0.018 to 0.148] | 0.142 [0.102 to 0.22] | 0.138 [0.111 to 0.376]
  Env-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Env-1-PTEg | 0.007 [0.004 to 0.013] | 0.057 [0.028 to 0.082] | 0.043 [0.033 to 0.099] | 0.093 [0.058 to 0.218] | 0.045 [0.036 to 0.12] | 0.033 [0.013 to 0.045] | 0.075 [0.033 to 0.119]
  Env-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Env-2-PTEg | 0.032 [0.012 to 0.033] | 0.036 [0.031 to 0.053] | 0.029 [0.016 to 0.068] | 0.057 [0.047 to 0.165] | 0.077 [0.01 to 0.083] | 0.032 [0.016 to 0.035] | 0.049 [0.032 to 0.066]
  Env-3-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Env-3-PTEg | 0.005 [-0.003 to 0.014] | 0.008 [0.008 to 0.044] | 0.025 [0.007 to 0.05] | 0.07 [0.032 to 0.139] | 0.031 [0.026 to 0.056] | 0.01 [0.005 to 0.04] | 0.037 [0.008 to 0.098]
  Gag-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Gag-1-PTEg | 0.06 [0.04 to 0.108] | 0.054 [0.035 to 0.062] | 0.163 [0.101 to 0.185] | 0.196 [0.053 to 0.272] | 0.015 [-0.001 to 0.031] | 0.108 [0.06 to 0.165] | 0.062 [0.048 to 0.211]
  Gag-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 9 | 10
  Gag-2-PTEg | 0.039 [0.001 to 0.058] | 0.011 [0.008 to 0.016] | 0.068 [0.059 to 0.089] | 0.134 [0.015 to 0.161] | 0.002 [-0.003 to 0.02] | 0.059 [0.039 to 0.071] | 0.017 [0.01 to 0.141]

19. Secondary Outcome: Occurrence of CD8+ T Cell Responses to the HIV Proteins Included in the Vaccine 2 Weeks After Each Boost
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. Response is positive if p<=0.00001. Data are excluded if the blood draw date was outside the visit window, the participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high. The responses at month 0.5 was not assayed.
Time Frame: Measured at Month 4.5
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Participants
  Any Env PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Any Env PTEg | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Any Gag PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Any Gag PTEg | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Any PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Any PTEg | 1 | 0 | 0 | 2 | 0 | 1 | 2
  Env-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Env-1-PTEg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Env-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Env-2-PTEg | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Env-3-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Env-3-PTEg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gag-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Gag-1-PTEg | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Gag-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Gag-2-PTEg | 1 | 0 | 0 | 0 | 0 | 1 | 0

20. Secondary Outcome: Level of CD8+ T Cell Responses to the HIV Proteins Included in the Vaccine 2 Weeks After Each Boost
Description: as for outcome 19
Time Frame: Measured at Month 4.5
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: % CD8+ T-cells
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
% CD8+ T-cells
  Any Env PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Any Env PTEg | 0.008 [-0.002 to 0.013] | 0.006 [-0.001 to 0.015] | 0.004 [0.003 to 0.018] | 0.015 [0.01 to 0.032] | 0.002 [-0.002 to 0.006] | 0.005 [0.003 to 0.013] | 0.01 [0.004 to 0.021]
  Any Gag PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Any Gag PTEg | 0.011 [0.006 to 0.124] | 0.006 [0 to 0.008] | 0.004 [0.001 to 0.014] | 0.005 [-0.001 to 0.025] | 0 [-0.009 to 0.012] | 0.006 [0.002 to 0.014] | 0.006 [-0.001 to 0.009]
  Any PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Any PTEg | 0.02 [0.018 to 0.122] | 0.009 [0.002 to 0.021] | 0.013 [0.007 to 0.037] | 0.031 [0.007 to 0.177] | 0.002 [-0.003 to 0.015] | 0.018 [0.008 to 0.037] | 0.02 [0.005 to 0.035]
  Env-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Env-1-PTEg | -0.003 [-0.003 to 0.013] | 0.001 [-0.008 to 0.007] | -0.005 [-0.007 to -0.003] | -0.002 [-0.005 to 0.003] | -0.005 [-0.009 to -0.005] | -0.003 [-0.007 to -0.003] | -0.002 [-0.005 to 0.003]
  Env-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Env-2-PTEg | 0.008 [-0.002 to 0.008] | 0.006 [-0.001 to 0.015] | 0.003 [-0.003 to 0.003] | 0.01 [0.004 to 0.019] | 0.002 [-0.002 to 0.006] | 0.003 [-0.002 to 0.008] | 0.01 [0.002 to 0.019]
  Env-3-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Env-3-PTEg | 0.004 [-0.005 to 0.007] | -0.002 [-0.005 to 0] | -0.003 [-0.006 to 0.005] | -0.001 [-0.002 to 0.02] | -0.005 [-0.007 to 0.002] | -0.003 [-0.005 to 0.005] | -0.001 [-0.004 to 0]
  Gag-1-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Gag-1-PTEg | 0.011 [0.006 to 0.124] | 0.006 [-0.002 to 0.008] | 0 [-0.003 to 0.002] | 0.004 [-0.001 to 0.025] | -0.001 [-0.009 to 0.002] | 0.002 [0 to 0.011] | 0.006 [-0.001 to 0.009]
  Gag-2-PTEg: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 9 | 10
  Gag-2-PTEg | 0.011 [-0.014 to 0.065] | -0.003 [-0.004 to 0] | 0 [-0.002 to 0.006] | 0.001 [-0.002 to 0.003] | -0.006 [-0.014 to 0.012] | 0.001 [-0.002 to 0.011] | -0.001 [-0.003 to 0.003]

21. Secondary Outcome: Occurrence of Env-specific IgG Responses for gp120, gp140, V1/V2, and the IDR of gp41 at 6 Months After the Final Boost
Description: as for outcome 9
Time Frame: Measured at Month 10
Population: "Overall Number of Participants Analyzed" includes the HIV uninfected participants with samples collected at the month 10 immunogenicity timepoint. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
Participants
  Con 6 gp120/B at Month 10: number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 5
  Con 6 gp120/B at Month 10 | 0 | 1 | 0 | 3 | 6 | 0 | 4
  Con S gp140 CFI at Month 10: number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 5
  Con S gp140 CFI at Month 10 | 2 | 2 | 4 | 3 | 7 | 6 | 5
  gp41 at Month 10: number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 5
  gp41 at Month 10 | 2 | 2 | 3 | 2 | 0 | 5 | 4
  gp70_B.CaseA_V1_V2 at Month 10: number analyzed (Participants) | 3 | 2 | 5 | 5 | 7 | 8 | 7
  gp70_B.CaseA_V1_V2 at Month 10 | 0 | 1 | 0 | 1 | 1 | 0 | 2

22. Secondary Outcome: Level of Env-specific IgG Responses for gp120, gp41, V1/V2, and the IDR of gp41 at 6 Months After the Final Boost
Description: as for outcome 9
Time Frame: Measured at Month 10
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost | Group 6: Boost | Group 7: Boost
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 10 | 10
fluorescence unit relative to background
  Con 6 gp120/B at Month 10: number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 5
  Con 6 gp120/B at Month 10 | 19 [1 to 37] | 443.5 [395.5 to 491.5] | 26.25 [15.5 to 57.25] | 2206.25 [718.25 to 3614.75] | 758.25 [325.25 to 1500] | 26.25 [11.75 to 37] | 718.25 [491.5 to 2206.25]
  Con S gp140 CFI at Month 10: number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 5
  Con S gp140 CFI at Month 10 | 6233.25 [3670 to 8796.5] | 5508 [3314.25 to 7701.75] | 9032.375 [6092.25 to 10348.375] | 13888.25 [13564.75 to 28461] | 8258.5 [2551.75 to 10231.25] | 8910 [3670 to 9041.25] | 13564.75 [7701.75 to 13888.25]
  gp41 at Month 10: number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 5
  gp41 at Month 10 | 7121.875 [3533 to 10710.75] | 15477.25 [4756.5 to 26198] | 9732 [3583.875 to 23070.625] | 14437.5 [2429 to 20424] | 492.5 [104.75 to 2117.75] | 7995.875 [3533 to 14183] | 14437.5 [4756.5 to 20424]
  gp70_B.CaseA_V1_V2 at Month 10: number analyzed (Participants) | 3 | 2 | 5 | 5 | 7 | 8 | 7
  gp70_B.CaseA_V1_V2 at Month 10 | 1 [1 to 44.75] | 132.875 [1 to 264.75] | 1 [1 to 1] | 14.25 [1 to 42.5] | 2.5 [1 to 69] | 1 [1 to 4.625] | 14.25 [1 to 264.75]

ADVERSE EVENTS:
Time Frame: Serious adverse events are collected throughout the study (months 0-10). Non-serious adverse events are collected through 30 days after each vaccination (at months 0 and 4).
Description: This table shows the number of participants reporting AEs by MedDRA preferred term and severity grade. The table was not grouped by the vaccine products because no vaccine related AE occurred.
Arm/Group | Group 1: Boost | Group 2: Boost | Group 3: Boost | Group 4: Boost | Group 5: Boost
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 2/4 | 4/4 | 3/6 | 2/6 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Boost (N=4) | Group 2: Boost (N=4) | Group 3: Boost (N=6) | Group 4: Boost (N=6) | Group 5: Boost (N=7)
Any Event in SOC (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Infections and infestations) | 1 (1) | 2 (7) | 2 (2) | 1 (1) | 3 (3)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT02852005/Prot_SAP_ICF_000.pdf